CLINICAL TRIAL: NCT05052060
Title: Effects of Pelvic Tilt Exercises With and Without Facet Joint Manipulation in Patients With Maigne's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/Lhr/0118 Aqsa Ashraf
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Back Pain
Keywords: Maigne's syndrome
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 19 patients will be treated with pelvic tilt exercises
  Interventions: Other: Group A
- Group B (Active Comparator): 19 patients will be treated with pelvic tilt exercises and facet joint manipulation.
  Interventions: Other: Group B

INTERVENTIONS:
Other: Group A — 19 patients will be treated with pelvic tilt exercises
  Arms: Group A
Other: Group B — 19 patients will be treated with pelvic tilt exercises and facet joint manipulation.
  Arms: Group B

SUMMARY:
The aim of this study is to find the effectiveness of exercise therapy and manipulative therapy for patients with maigne's syndrome. It is a Randomized clinical trial and convenient random sampling is to be used with an inclusion criteria of patients having maignes syndrome without having neurological signs and specific spinal pathology like disc lesion ,malignancy or inflammatory disease and any other major medical conditions .

DETAILED DESCRIPTION:
Maigne's syndrome is a pain disorder of low back which mainly affects the thoracolumbar junction of spine ,normally called as thoracolumber junction syndrome.It eludes healthcare professinals because of its pain presentation ,which is far away from the problematic site .Dr.Maigne wo was the founder of this syndrome stated that ,the most important cause behind this syndrome is Intervertebral dysfynction.It causes irritation ,inflammation and mild degeneration of involved intervertebral structures .Referred pain is the most important chracteristic of this syndrome which mainly involves lower back region ,groin ,lumbosacral region ,lower abdominl region and SI joint .Diagnostic criteria is based on 4 principles which need keen observation because many professionals simply fail to recognize it .

To treat the Maigne's syndrome manipulation and exercise therapy is directed. In exercise therapy pelvic tilt exercises which include simple pelvic tilt ,addition of pelvic muscles ,addition of back extension with pelvic tilt and positioning of hands on back while performing exercise .and on the other hand in manipulative therapy facet joint manipulation included to reduce the pain , to increase pain free movement and to decrease other associated sign and symptoms.

The aim of this study is to find the effectiveness of exercise therapy and manipulative therapy for patients with maigne's syndrome. It is a Randomized clinical trial and convenient random sampling is to be used with an inclusion criteria of patients having maignes syndrome without having neurological signs and specific spinal pathology like disc lesion ,malignancy or inflammatory disease and any other major medical conditions .patients also having lumbar flattening in lumbar lordosis according to MRI will be excluded.The main purpose of this randomized clinical trial will be to find out the effects of pelvic tilt exercises with and without facet joint manipulation in reducing pain and improvement in pain free sitting in patients with maigne's syndrome. Patients will be randomly allocated into two groups, Group A will receive exercise therapy intervention and Group B will receive manipulative therapy. Total duration of study will be three months with assessment will be done before treatment and after every 4 weeks. Numeric pain rating scale and oswestry index will be used to measure the outcomes. After collecting data from defined study setting, data will be entered and analyzed by using Statistical Package for the Social Sciences (SPSS) for Windows software, version 25. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages ranging between 20-40 years among male
* Eligibility criteria include:
* Tenderness on palpation test at thoracolumbar junction
* Sensitivity difference on illiac crest
* Positive skin rounding test
* patients must have nonspecific unilateral pain in the lower lateral region of spine and radiates along the pelvis into the pubic region
* Written informed voluntary consent

Exclusion Criteria:

* Participants will be excluded if they had:
* specific spinal pathology (e.g. disc lesions, malignancy, or inflammatory disease) or any other major medical pathology.
* Patients having flattening in the lumbar lordosis according to the lumbar MRI results were excluded

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Numeric Pain rating Scale | 6 weeks
  To measure pain, Numeric Pain Rating Scale (NPRS) is anchored by terms describing pain severity extremes. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Modified Oswestry index | 6 weeks
  to measure disability, The Modified Oswestry disability index (MODI) has been developed to assess pain related disability. The questionnaire consists of 10 items addressing different aspects of function. Each item is scored from 0 to 5, with higher values representing greater disability. The total score is multiplied by 2 and expressed as a percentage

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- General Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SR, Lee MJ, Lee SJ, Suh YS, Kim DH, Hong JH. Thoracolumbar Junction Syndrome Causing Pain around Posterior Iliac Crest: A Case Report. Korean J Fam Med. 2013 Mar;34(2):152-5. doi: 10.4082/kjfm.2013.34.2.152. Epub 2013 Mar 20. PMID 23560215
- [Background] Maigne R. Pain Syndromes of the Thoracolumbar Junction: A Frequent Source of Misdiagnosis. Physical Medicine and Rehabilitation Clinics Of North America. 1997;8(1):87-100.
- [Background] Aktas I, Palamar D, Ozkan FU, Akgun K. Testicular pain due to thoracolumbar junction syndrome: a case report. Revista Internacional de Andrología. 2016;14(4):148-52.